CLINICAL TRIAL: NCT05244005
Title: Incidence, Risk Factors and Outcomes for Early and Delayed Extubatiion Failure in Critically Ill Cirrhotic Patients
Brief Title: Extubation Failure in Critically Ill Cirrhotic Patients.
Acronym: FREELIVER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0731
Record Dates: First submitted 2022-01-10; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Cirrhosis; Mechanical Ventilation Complication; Critical Illness
Keywords: Extubation failure; Mechanical ventilation; Risk factors
MeSH Terms: conditions — Fibrosis; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Although a life-saving intervention, invasive mechanical ventilation (MV) prone to complications and side effects.

Cirrhotic patients with a need of prolonged MV have a poor prognosis in ICU compared to general population of critically ill patients. The optimal time for weaning from MV and extubation is therefore a crucial objective. Extubation failure is defined as the need for reintubation within 48-72 hours (early). This time frame is sometimes extended to 7 days (delayed), especially when noninvasive ventilation is used during extubation (SFAR-SRLF 2018 recommendations). Some studies have investigated the risk factors for extubation failure in general population of critically ill patients, and in some specific subpopulations (COPD, brain injury, elderly). But little is known about extubation failure in cirrhotic patients admitted in ICU.

The aim of the present study is to describe the incidence and identify specific risk factors for extubation failure in cirrhotic critically ill patients. Ultrasound and clinical data will be collected and analysed during the ICU stay.

DETAILED DESCRIPTION:
Mechanical ventilation (MV) is a life saving therapy for many critically ill patients. However, it is associated with major complications (ventilator-associated pneumonia, resuscitation neuromyopathy, etc.) that affect the prognosis. The optimal time for weaning from MV and extubation is therefore a major question. The decision to extubate is usually made as soon as the patient meets predefined weaning criteria and succed a spontaneous breathing test (SBT). However, extubation failure occurs in 10 to 20% of patients who suceeded an SBT in general critically ill patients. Extubation failure is defined as the need for reintubation within 48-72 hours. This time frame is sometimes extended to 7 days, especially when noninvasive ventilation is used during extubation (SFAR-SRLF 2018 recommendations). Early and delayed extubation Failure are then defines as failure within 48 hours and between day 2 and day 7 respectively. The decision to extubate in even more challenging because failure is associated with an overall increase in the duration of MV, an increased need for tracheostomy, higher medical costs but also particularly higher mortality. There is also evidence that extubation failure is not only a marker of more severe disease, but independently affects patient survival, regardless of the severity of the underlying disease.

Cirrhotic patients represent 5 to 8% of all ICU admissions. Their mortality is significantly higher than the general population (34 to 69% depending on the reason for admission). The need for MV is one of the main causes of admission of cirrhotic patients to the ICU, but it is also one of their main risk factors for mortality (60 to 91% for MV cirhhotic patients in ICU). The proportion of cirrhotic patients admitted to the ICU is constantly increasing due to the improvement of the global prognosis linked to novel therapies (transjugular intrahepatic porto-systemic shunt, liver dialysis, liver transplantation). Numerous studies have investigated the risk factors for extubation failure in critically ill patients. The largest multicenter cohort (FREE-REA study, sponsor CHU of Montpellier, first author Pr Samir Jaber, PMCID: PMC6151191), included 11% of cirrhotic patients out of 1453 patients in total. A post-hoc analysis of these data showed similar incidences of extubation failure at H48 between cirrhotic and non-cirrhotic patients (10.5% Vs 9.1%; p=0.57) but a higher incidence of delayed extubation failure (at D7) in cirrhotic patients (18.9% Vs 11.5%; p<0.01). However, the specific causes and risk factors were not clearly identified, and no study to date has specifically looked at this population and its risk factors for extubation failure.

The aim of the present study is to describe the incidence and identify specific risk factors for extubation failure in cirrhotic critically ill patients. Ultrasound and clinical data will be collected and analysed during the ICU stay

ELIGIBILITY:
Inclusion criteria:

* Adult patients
* Known history of cirrhosis or diagnosis of cirrhosis during the ICU stay
* Invasive mechanical ventilation for more than 6 hours
* Eligible for extubation according to the physician in charge

Exclusion criteria:

* Pregnancy,
* Age below 18
* Terminal extubation
* Absence of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive critically ill patients admitted to the intensive care unit of Saint Eloi University teaching hospital with a history or diagnosis of cirrhosis and requiring invasive mechanical ventilation for more than 6 hours.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of extubation failure | From extubation (day 0) to day 7 after extubation
  Incidence of extubation failure in cirrhotic patients ventilated for more than 6 hours in the ICU

SECONDARY OUTCOMES:
Risk factors for extubation failure | From extubation (day 0) to day 7 after extubation
  Risk factors for extubation failure

CONTACTS AND LOCATIONS:
Overall Officials: Yassir AARAB, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC